CLINICAL TRIAL: NCT00414310
Title: Phase II Randomized Study of Low-Dose Decitabine (5-AZA-2'-Deoxycytidine) With or Without Valproic Acid in Myelodysplastic Syndrome (MDS) and Acute Myelogenous Leukemia -"SPORE"
Brief Title: Decitabine (DAC) w/ or w/o Valproic Acid (VPA) in Myelodysplastic Syndrome (MDS) and Acute Myelogenous Leukemia (AML)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0686; NCI-2012-01396 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2006-12-19; First posted 2006-12-21 (Estimated); Results first posted 2015-08-13 (Estimated); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Myelodysplastic Syndrome; Acute Myelogenous Leukemia
Keywords: Decitabine; Dacogen; 5-AZA; Valproic Acid; Myelodysplastic Syndrome; Acute Myelogenous Leukemia; MDS; AML
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — Decitabine; Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Decitabine (Experimental): Decitabine 20 mg/m^2 intravenous (IV) over 1 hour daily for 5 days.
  Interventions: Drug: Decitabine
- Decitabine + Valproic Acid (Experimental): Decitabine 20 mg/m^2 intravenous (IV) over 1 hour daily for 5 days. Valproic Acid 50 mg/kg orally daily for 7 days.
  Interventions: Drug: Decitabine; Drug: Valproic Acid

INTERVENTIONS:
Drug: Decitabine — 20 mg/m^2 IV over 1 hour daily for 5 days.
  Other Names: Dacogen
Drug: Valproic Acid — 50 mg/kg orally daily for 7 days
  Arms: Decitabine + Valproic Acid

SUMMARY:
The goal of this clinical research study is to find out if decitabine, given with or without valproic acid, can help to control AML or MDS. The safety of both treatments will also be studied.

DETAILED DESCRIPTION:
Decitabine and valproic acid are both designed to cause changes in different groups of proteins that are attached to DNA (the genetic material of cells), which may cause cancer cells to die. Researchers want to see if a combination of valproic acid with decitabine can help improve disease response as well as how long responses last in treating MDS and AML.

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the toss of a coin) to 1 of 2 groups. Participants in one group will receive decitabine. Participants in the other group will receive decitabine and valproic acid. You will have an equal chance of being assigned to either group at first. After 20 participants are enrolled in each group, you will have a greater chance of being assigned to the group that is showing better results.

Participants in both groups will receive decitabine on Day 1 through a central venous catheter (CVC) in a vein over 1 hour each day for 5 days. A central venous catheter is a sterile flexible tube that will be placed into a large vein while you are under local anesthesia. Your doctor will explain this procedure to you in more detail, and you will be required to sign a separate consent form for this procedure. Participants who are assigned to also get valproic acid will take the drug by mouth on Days 1-7 (7 days in a row).

On Day 0 (the day before treatment begins) or on Day 1, you will have a physical exam, including measurement of your vital signs. Blood (about 2 teaspoons) will be drawn on or about Days 0 or 1, 5, and 10 (if your routine blood tests were found to be abnormal) to learn the status of the disease.

Routine blood draws (about 4 teaspoons) will be done 1-2 times weekly for the first cycle and then every 2-4 weeks in further cycles. You will have another bone marrow aspiration to check disease response to treatment, and then you will have one every 1-3 cycles. One (1) cycle of treatment is 4-8 weeks long.

You may remain on this study as long as you are benefitting or up to 2 years after you first achieve a complete response. Your dose level may be decreased depending on the side effects you may experience. However, if the disease gets worse or you experience any intolerable side effects, you will be taken off this study.

This is an investigational study. Decitabine is FDA approved and commercially available for the treatment of MDS. Valproic acid is FDA approved and commercially available for the treatment of seizure disorders. Up to 150 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with MDS and > 5% blasts or IPSS risk intermediate or high; patients with CMML; patients with AML who are age 60 or older. No prior intensive chemotherapy or high-dose ara-C (> 1g/m2). No prior azacytidine for 3 cycles or more or prior decitabine for 2 cycles or more. Prior biologic therapies, targeted therapies, or single agent chemotherapy allowed.Patients must have been off chemotherapy for 2 weeks prior to entering this study and recovered from the toxic effects of that therapy, unless there is evidence of rapidly progressive disease.
2. Continued from #1: Hydroxyurea is permitted for control of counts prior to treatment. Procrit, granulocyte colony-stimulating factor (GCSF) are allowed before therapy. Procrit, GCSF or other growth factors are permitted on therapy. Use of hydroxyurea with rapidly proliferative disease is allowed for the first two weeks on therapy.
3. Performance 0-2 (ECOG). Adequate liver function (bilirubin of < 2mg/dl) and renal function (creatinine < 2mg/dl). Adequate cardiac functions (NYHA cardiac III-IV excluded). ALT < 2.5x institutional upper limit of normal.
4. Signed informed consent.

Exclusion Criteria:

1. Nursing and pregnant females. Patients of childbearing potential should practice effective methods of contraception. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
2. Active and uncontrolled infections.
3. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements.
4. Known ornithine transcarbamylase disorder.
5. Patients requiring continuous valproic acid treatment for the control of seizure disorders.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2006-12; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hagop Kantarjian, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 12/13/2006 to 07/05/2010. All recruitment done at The University of Texas MD Anderson Cancer Center.
Pre-assignment Details: Of the 153 participants registered on the study for Decitabine (DAC) with or without Valproic Acid (VPA) in Myelodysplastic Syndrome (MDS) and Acute Myelogenous Leukemia (AML), three were screen failures therefore 150 patients were randomized with 149 participants treated.
Groups:
- Decitabine + Valproic Acid: Decitabine 20 mg/m^2 IV over 1 hour daily for 5 days. Valproic Acid 50 mg/kg orally daily for 7 days.
Period: Overall Study
Arm/Group | Decitabine | Decitabine + Valproic Acid
Started | 71 | 79
Completed | 70 | 79
Not Completed | 1 | 0
Not completed — Not treated | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Decitabine | Decitabine + Valproic Acid | Total
Number analyzed (Participants) | 71 | 79 | 150
Age, Continuous [Median (Full Range); unit: years] | 71 [39 to 85] | 66 [20 to 90] | 69 [20 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 37 | 58
  Male | 50 | 42 | 92
Region of Enrollment [Number; unit: participants]
  United States | 71 | 79 | 150

OUTCOME MEASURES:

1. Primary Outcome: Participant Response Rates to Decitabine With or Without Valproic Acid in MDS and AML
Description: Complete Remission (CR): CR defined as normalization of peripheral blood and bone marrow with < 5% bone marrow blasts, a peripheral blood granulocyte count > (1.0 x 10^9/ L, and a platelet count > 100 x 10^9/L). CRi or complete remission with incomplete platelet recovery is defined as above, but platelets <100 x 109/L. Partial Remission: as above except for the presence of 6-15% marrow blasts, or 50% reduction if <15% at start of treatment. Clinical Benefit: In MDS/CMML, as per International Working Group (IWG) criteria, platelets increase by 50% and to above 30 x 10^9/L untransfused (if lower than that pretherapy); or granulocytes increase by 100% and to above 10^9/L (if lower than that pretherapy); or hemoglobin increase by 2 g/dl; or transfusion independent; or splenomegaly reduction by > 50%; or monocytosis reduction by > 50% if pretreatment > 5 x 10^9/L. In addition to IWG criteria, in AML, a decrease in bone marrow blasts to <5% also considered clinical benefit.
Time Frame: 1 Year
Population: One enrolled participant on the Decitabine arm was not treated, therefore not evaluable for response.
Measure: Number; unit: Percentage of Participants
Arm/Group | Decitabine | Decitabine + Valproic Acid
Number analyzed (Participants) | 70 | 79
Percentage of Participants
  Complete Remission (CR) | 22 | 29
  Complete Remission Without Platelet Recovery (CRi) | 6 | 9
  Partial Remission (PD) | 0 | 1

2. Secondary Outcome: Response Duration
Description: The date of Response to the date of loss of response or last follow-up.
Time Frame: Up to 60 months
Population: One enrolled participant on the Decitabine arm was not treated, therefore not evaluable for response.
Measure: Median (Full Range); unit: Months
Arm/Group | Decitabine | Decitabine + Valproic Acid
Number analyzed (Participants) | 70 | 79
Months | 12.9 [1 to 55] | 6.3 [2 to 57]

3. Secondary Outcome: Overall Survival Rate
Description: Time from date of treatment start until date of death due to any cause or last Follow-up.
Time Frame: Up to 7 years
Population: One enrolled participant on the Decitabine arm was not treated, therefore not evaluable for response.
Measure: Median (Full Range); unit: months
Arm/Group | Decitabine | Decitabine + Valproic Acid
Number analyzed (Participants) | 70 | 79
months | 11.2 [0 to 70] | 11.9 [0 to 73]

ADVERSE EVENTS:
Time Frame: Adverse events reported during each treatment course every 4-8 weeks and extending 30 days beyond the last day of active treatment. Overall period: 12/2006 to 07/2011.
Arm/Group | Decitabine | Decitabine + Valproic Acid
Serious Adverse Events (participants affected / at risk) | 43/71 | 49/79
Other Adverse Events (participants affected / at risk) | 27/71 | 36/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Decitabine (N=71) | Decitabine + Valproic Acid (N=79)
Edema (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Gastrointestinal Hemorrhage (Blood and lymphatic system disorders) | 3 (4) | 0 (0)
Hemorrhage (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
bilateral deviationn eye (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Arrhythmia (Cardiac disorders) | 2 (2) | 2 (2)
cardiac hypotension (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac infarction (Cardiac disorders) | 0 (0) | 1 (1)
Congestive Heart Failure (Cardiac disorders) | 2 (2) | 3 (3)
Hypotension (Cardiac disorders) | 2 (2) | 0 (0)
Left ventricular diastolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 2 (2) | 0 (0)
Pacemaker malfuncion (Cardiac disorders) | 0 (0) | 1 (1)
Pulmonary hypertension (Cardiac disorders) | 0 (0) | 1 (1)
Pulmonary Obstruction (Cardiac disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea and Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Back Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death (Gastrointestinal disorders) | 9 (9) | 5 (5)
Epigastric pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fall (Gastrointestinal disorders) | 2 (2) | 0 (0)
Fatigue (Gastrointestinal disorders) | 1 (1) | 0 (0)
fever (Gastrointestinal disorders) | 0 (0) | 3 (3)
Joint pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tumor lysis syndrome (Gastrointestinal disorders) | 0 (0) | 2 (2)
Weakness (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bacteremia (Infections and infestations) | 1 (1) | 4 (4)
Infection other (Infections and infestations) | 10 (16) | 9 (9)
Neutropenic Fever (Infections and infestations) | 11 (13) | 22 (34)
Pancreatitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 10 (10) | 11 (13)
Altered Mental Status (Nervous system disorders) | 1 (1) | 1 (2)
Anxiety and Depression (Nervous system disorders) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Confusion (Nervous system disorders) | 1 (1) | 0 (0)
encephalopathy (Nervous system disorders) | 0 (0) | 1 (2)
Hallucinations (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 4 (4)
Stroke (Nervous system disorders) | 2 (2) | 1 (1)
visual loss (Nervous system disorders) | 1 (1) | 0 (0)
acute renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | 1 (1) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
cholecystectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 2 (2)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Decitabine (N=71) | Decitabine + Valproic Acid (N=79)
Edema: limb (Blood and lymphatic system disorders) | 1 (1) | 1 (2)
Edema: trunk/genital (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardiac Arrhythmia (Cardiac disorders) | 2 (2) | 2 (2)
Cardiac General (Cardiac disorders) | 1 (1) | 1 (1)
Vision-blurred vision (Eye disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 4 (4)
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis/stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 10 (12)
Fatigue (General disorders) | 6 (6) | 9 (9)
Pain (General disorders) | 3 (3) | 2 (2)
Cholecystitis (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 8 (10) | 8 (11)
Neutropenic Fever (Infections and infestations) | 10 (13) | 12 (17)
Opportunistic infection (Infections and infestations) | 2 (2) | 3 (3)
Creatinine (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
hyperbilirubinemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Metabolic/Laboratory-Other (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
CNS cerebrovascular ischemia (Nervous system disorders) | 0 (0) | 1 (1)
Confusion (Nervous system disorders) | 1 (1) | 3 (3)
Dizziness (Nervous system disorders) | 0 (0) | 5 (5)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (2)
Mood alteration (Nervous system disorders) | 0 (0) | 1 (1)
Neurology Other (Nervous system disorders) | 0 (0) | 4 (4)
Sensory Neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 6 (7)
Renal Failure (Renal and urinary disorders) | 4 (4) | 1 (1)
Renal Gentitourinary other (Renal and urinary disorders) | 0 (0) | 1 (1)
Adult Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary/Upper Respiratory-Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatology/Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes